CLINICAL TRIAL: NCT06793384
Title: Applying Cognitive Stimulation Therapy (CST) and Virtual Reality-based CST on People with Concurrent Visual Impairment and Dementia: a Feasibility Pilot Study
Brief Title: Virtual Reality in Cognitive Stimulation Therapy for Visually Impaired Older Individuals with Dementia
Acronym: VR-CST-PwDVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other); The Hong Kong Society for the Blind (Unknown); Tung Wah College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA240610
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Dementia Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional CST group (Active Comparator): A total 14 sessions of conventional cognitive stimulation therapy (CST) with different themes were delivered twice a week to patients with dementia in groups of four to five. Therapy materials included real objects, pictures and videos presented via iPADs where users can enlarge the images manually or under facilitator's assistancd.
  Interventions: Behavioral: Conventional Cognitive Stimulation Therapy (Conventional CST)
- VR-CST (Experimental): A total of 14 sessions of virtual reality cognitive stimulation therapy (VR-CST) with different themes were delivered twice a week to patients with dementia in groups of four to five. In the VR-CST condition, participants wore a head-mounted display (HMD; model: DPVR P1 Pro Headset) for the themed activities in every session except sessions 1 and 14. In these two sessions, group physical activities (such as passing a ball from one participant to another) were conducted, so no HMDs were used. In other sessions, panoramic images (e.g., wet market) and videos (e.g., the neighborhood surroundings) prepared by the project team were mainly used, supplemented by 2-dimensional images /videos in which preparing panoramic images/videos was deemed impossible.
  Interventions: Behavioral: Virtual reality based Cognitive Stimulation Therapy (VR-CST)

INTERVENTIONS:
Behavioral: Virtual reality based Cognitive Stimulation Therapy (VR-CST) — In the VR-CST condition, participants wore a head-mounted display (HMD; model: DPVR P1 Pro Headset) for the themed activities in every session except sessions 1 and 14. In these two sessions, group physical activities (such as passing a ball from one participant to another) were conducted, so no HMDs were used. In other sessions, panoramic images (e.g., wet market) and videos (e.g., the neighborhood surroundings) prepared by the project team were mainly used, supplemented by 2-dimensional images /videos in which preparing panoramic images/videos was deemed impossible. Such a situation occurred in Session 5 (current affairs), in which news clips or captions from newspaper websites served as more appropriate content for discussion than self-created panoramic images/videos.
  Arms: VR-CST
Behavioral: Conventional Cognitive Stimulation Therapy (Conventional CST) — In the conventional CST group, 2-dimensional images/videos illustrating content identical to the VR-CST condition were displayed via tablet computers (see Table 2 for details) in which participants could manipulate the size of the image depicted or the pace of the videos with the help of the facilitator/therapy assistant.
  Arms: Conventional CST group

SUMMARY:
Both visual impairment and dementia are prevalent in the elderly population. Cognitive stimulation therapy (CST) is an evidence-based intervention for people with mild-to-moderate dementia. Virtual reality (VR) has been used in cognitive rehabilitation. However, the efficacy of CST and the feasibility of incorporating VR into therapy targeting people with dementia and visual impairment (PwDVI) have rarely been explored. The current pilot study addressed two issues: 1) To study the efficacy of conventional CST on PwDVI in different cognitive domains and 2) To explore the feasibility and efficacy of VR-CST on PwDVI in various cognitive domains.

ELIGIBILITY:
Inclusion Criteria:

1. Cantonese speakers;
2. suspected or having a medical diagnosis of dementia, with the Montreal Cognitive Assessment 5-minute protocol (MoCA-5) score ranging from 2 to 17, which is equal to the Cantonese Mini Mental State Examination (MMSE) score ranging from 10 to 24 by using the conversion table from Wong et al,
3. a diagnosis of mild to moderate visual impairment determined by an optometrist,
4. no other disability including physical illness, learning disability and severe hearing impairment that may affect participation in group activity,
5. not currently on psychiatric medication/cognitive intervention, (6) no history of other neurological diseases, and

(7) did not receive any prior CST.

Exclusion Criteria:

1. currently on psychiatric medication/cognitive intervention, (6) no history of other neurological diseases,
2. currently on psychiatric medication/cognitive intervention, (6) no history of other neurological diseases,
3. prior exposure to CST

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
The Hong Kong version of the Montreal Cognitive Assessment for the Visually Impaired (HKMoCA-VI) | The assessment was administered three times 15 days before and after treatment.
  It is a standarized assessment for global cognition for people with visual impairment.

SECONDARY OUTCOMES:
Holden Communication Scale | It was administered once one week before and after the intervention.
  It is a questionnaire to evaluate the participants' communication and social behavior from a caregiver's perspective. Ratings were given by the formal carers of the old age homes for the visually imapired.
Cantonese version of the Amsterdam-Nijmegan Everyday Language Test (CANELT) | Three times 15 days before and after treatment
  The test portrays 20 real-life situations encompassing different communicative functions, was conducted to evaluate functional communication quantitively. Scores were given based on the accuracy and completeness of the main concepts produced by the subjects.
Procedural description of making a ham-and-egg sandwich | The assessment was administered three times 15 days before and after treatment.
  A picture depicting a loaf of bread, ham and an egg were presented to the subject and s/he will be asked to describe the procedures of making an egg-and-ham sandwich as detailed as possible.
Synonym judgement | The assessment was administered three times 15 days before and after treatment.
  A pair of words were presented auditorily and the participants were asked to judge if the pair of words were synonymous or not.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Society for the Blind, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Participants' performance (raw scores) on primary and secondary outcomes throughout the study period will be shared on an open access repository (e.g., OSF).
Supporting Information: ICF
Time Frame: From Feb 2025 to Jan 2034
Access Criteria: There is no restriction to access.